CLINICAL TRIAL: NCT06071078
Title: Impact of a Protocol for Announcing the Limitation and Discontinuation of Therapies in the Emergency Departments on the Stress of Families
Brief Title: Impact of a Protocol for Announcing Decision of Withholding and Withdrawing Life-sustaining Treatments on the Stress of the Relatives in the Emergency Departments
Acronym: DISCUSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69HCL20_0070
Record Dates: First submitted 2023-08-08; First posted 2023-10-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: End of Life
Keywords: Limitation and cessation of treatment; Stress; End of life
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: Stepped-wedge trial
Who Masked: Outcomes Assessor
Masking Description: The evaluation will be carried out centrally for all the subjects included, 90 days after the announcement to the emergency room, by a psychologist, trained in the data collection interview, on the telephone, without the knowledge of the group (training provided or not to caregivers).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DISCUSS announcement protocol (Experimental): Model protocol for announcing decision of withholding and withdrawing life-sustaining treatments, with human simulation and the intervention of partner families in a simulation center and in situ, on the reduction of family stress following the announcement of a decision of withholding and withdrawing life-sustaining treatments in the emergency departments
  Interventions: Behavioral: Training of professionals according to the DISCUSS announcement protocol
- Control (No Intervention): Individuals will receive the usual practices.

INTERVENTIONS:
Behavioral: Training of professionals according to the DISCUSS announcement protocol — The emergency services will be divided into 4 clusters (2 or 3 services per cluster). Each cluster will belong successively to the control arm and then to the intervention arm according to a 5 successive steps of 4 months duration (stepped wedge method). The deployment of the training will therefore not be done simultaneously in the different services.
  Individuals in this group will have received a decision of withholding and withdrawing life-sustaining treatments according to the DISCUSS announcement protocol, by a professional trained in this procedure.
  Arms: DISCUSS announcement protocol

SUMMARY:
Death is a daily reality in the emergency department. Deaths represent 0.3 to 0.5% of emergency admissions, i.e. approximately 26,000 per year for the whole of France. For 80% of these deceased patients, a decision of withholding and withdrawing life-sustaining treatments was made in the emergency departments. The announcement of death and decision of withholding and withdrawing life-sustaining treatments in this context is complex because of the lack of time and the inappropriate places for the announcement. In addition, the short delay in the occurrence of these events may increase the stress and anxiety of families who are unprepared for the announcement. However, there is little data in the literature on the impact on families in terms of their experience of announcements in the emergency context.

It has been established that symptoms of anxiety and depression are correlated with the onset of posttraumatic stress disorder and that the latter is more important in the families of deceased patients and after a decision to undergo decision of withholding and withdrawing life-sustaining treatments in the intensive care unit. In order to identify it, several tools have been developed, including the Impact Event Scale (IES), which has been widely used to detect symptoms related to PTSD.

It has also been shown that training nursing staff in communication skills or the use of written support in dealing with the families of patients who have died in intensive care reduces the appearance of post-traumatic stress symptoms.

Human simulation is a pedagogical technique for learning interpersonal skills through role playing. It is used, among other things, in announcement situations in medicine. Nevertheless, its impact in emergency medicine has not been evaluated.

Moreover, it has been shown that the involvement of the patient-partner in the care process must be improved and encouraged and that its impact has yet to be evaluated. Therefore, the objective is to evaluate the impact of a model protocol for announcing decision of withholding and withdrawing life-sustaining treatments, with human simulation and the intervention of partner families in a simulation center and in situ, on the reduction of family stress following the announcement of a decision of withholding and withdrawing life-sustaining treatments in the emergency departments.

Hypothesis is that training all emergency department caregivers in the use of a model announcement protocol with the support of human simulation, combining training of pairs in a simulation center and in situ training, and the participation of partner families, would allow for a better understanding of announce of withholding and withdrawing life-sustaining treatments decision in the emergency department and reduce their impact on families in terms of the occurrence of acute stress and post-traumatic stress symptoms.

ELIGIBILITY:
Inclusion Criteria:

For relatives, will be included in the study:

* Trusted persons, families or relatives present in the emergency departments and to whom the 1st announcement of a decision to limit or stop therapies is made by a physician participating in the study. Several persons can be included for the same patient (maximum 3) in the following order: trusted person > family > close relative.
* Age of trusted person, family or close friends over 18 years old.
* Informed consent given and voice rights signed for families accepting the semi-directed interview.

For caregivers, also included in the study will be:

* Caregivers on participating wards.
* Informed consent given and voice rights signed for families accepting the semi-directed interview.

For partner families, will be included in the study:

* Trusted persons, families or relatives present in the emergency department and to whom the 1st announcement of a decision to limit or stop therapy by a physician in a participating emergency department is made.
* Age of trusted person, family or close friends over 18 years old.
* Signed consent for the right to voice recording.

Exclusion Criteria:

For relatives:

* Trusted person, family or close friend whose announcement would have been made entirely by telephone.
* Trusted person, family or close friend unable to understand or write in French.
* Pregnant women, women in labor or nursing mothers.
* Persons deprived of liberty by a judicial or administrative decision.
* Persons under psychiatric care.
* Persons admitted to a health or social institution for purposes other than research.
* Persons of full age who are subjects to a legal protection measure (guardians, curators).
* Persons not affiliated to a social security system or beneficiaries of a similar system.

For caregivers:

- Persons not affiliated to a social security system or beneficiaries of a similar system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Assessment of post-traumatic stress symptoms | Day 90 after the announcement in the emergency department
  Post-traumatic stress symptoms will be assessed using IES (Impact of Even Scale) at 90 days. The IES score is composed of 15 questions. The maximum score is 75, the minimum score is 0. A high score reflects an improvement/worsening of the condition of the subject participating in the study. This evaluation will be conducted by a psychologist, trained in the data collection interview, on the telephone, unbeknownst to the group (training given or not to the caregiver).

SECONDARY OUTCOMES:
Families - Effect of the protocol for announcing limitations or cessation of treatment - Post-traumatic stress symptoms | Day 7 after the announcement in the emergency department
  Post-traumatic symptoms will be assessed using the Impact of Event Scale (IES) at 7 days. The IES score is composed of 15 questions. The maximum score is 75, the minimum score is 0. A high score reflects a worsening of the condition of the subject participating in the study.
Families - Effect of the protocol for announcing limitations or cessation of treatment - Post-traumatic stress symptoms | Day 30 after the announcement in the emergency department
  Post-traumatic symptoms will be assessed using the Impact of Event Scale (IES) at 30 days. The IES score is composed of 15 questions. The maximum score is 75, the minimum score is 0. A high score reflects a worsening of the condition of the subject participating in the study.
Families - Effect of the protocol for announcing therapeutic limitations or cessation - Diagnosis of post-traumatic stress | Day 90 after the announcement in the emergency department
  The diagnosis of post-traumatic stress at 90 days will be established by the PCL-5 (Post Traumatic Stress Disorder Checklist for DSM-5, "Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition"). The PCL-5 scale is composed of 20 items. The maximum score is 80, the minimum score is 0. A high score reflects a worsening of the condition of the subject participating in the study.
Families - Effect of the protocol for announcing therapeutic limitations or cessation - Anxiety and depression symptoms | Day 7 after the announcement in the emergency department
  Anxiety and depression symptoms will be assessed using the HADS (Hospital Anxiety and Depression Scale) score at 7 days. The HADS score is composed of 14 items. The maximum score for the anxiety part is 21 and for the depression part is 21, the minimum score is 0. A high score reflects a worsening of the condition of the subject participating in the study.
Families - Effect of the protocol for announcing therapeutic limitations or cessation - Anxiety and depression symptoms | Day 30 after the announcement in the emergency department
  Anxiety and depression symptoms will be assessed using the HADS (Hospital Anxiety and Depression Scale) score at 30 days. The HADS score is composed of 14 items. The maximum score for the anxiety part is 21 and for the depression part is 21, the minimum score is 0. A high score reflects a worsening of the condition of the subject participating in the study.
Families - Effect of the protocol for announcing therapeutic limitations or cessation - Anxiety and depression symptoms | Day 90 after the announcement in the emergency department
  Anxiety and depression symptoms will be assessed using the HADS (Hospital Anxiety and Depression Scale) score at 90 days. The HADS score is composed of 14 items. The maximum score for the anxiety part is 21 and for the depression part is 21, the minimum score is 0. A high score reflects a worsening of the condition of the subject participating in the study.
Families - Effect of the protocol for announcing therapeutic limitations or cessation - Families' experiences | Day 7 after the announcement in the emergency department
  The experience of the relatives will be evaluated through questions collected 7 days after the announcement by a psychologist (questions on experience and feelings).
Families - Effect of the protocol for announcing therapeutic limitations or cessation - Families' experiences in the training group | Day 90 after the announcement in the emergency department
  The experiences of the families will be evaluated on a sample of the families in this "training" group. To do so, a psychologist with these families will conduct semi-directive interviews.
Families - Effect of the protocol for announcing therapeutic limitations or cessation - Impact on the socio-professional life of families | Day 90 after the announcement in the emergency department
  The impact of the announcement on the socio-professional life of families will be assessed by the presence of at least one work stoppage related to a visit to the emergency department within 90 days of the announcement, followed by the number of days of work stoppage. These data will be collected during the 90-day telephone interview with the psychologist.
Caregivers - Satisfaction with protocol training | Month 4, Month 8, Month 12, Month 16, Month 20 after training
  Caregivers' satisfaction will be assessed using a self-questionnaire based on the model recommended by the French National Authority for Health (Haute Autorité de Santé) and used in the SAMSEI program ("Stratégies d'Apprentissage des Métiers de Santé en Environnement Immersif", or "Learning Strategies for Healthcare Professions in an Immersive Environment" in English) and the Lyon Sud Health Simulation Center. The questionnaire will be completed by participants at the end of protocol training. The questionnaire will assess interest, practical usefulness, density of information, compliance with objectives, material conditions of training, participant activity and motivation to continue training.
Caregivers - Impact of partner families' involvement in training on professionals | Month 4, Month 8, Month 12, Month 16, Month 20 before training
  Caregivers' views on the involvement of partner families will be assessed by means of a self-administered questionnaire and during semi-structured interviews. The questionnaire will be completed by the participants before and after the training and intervention of the partner families.
Caregivers - Evaluating assertiveness at the communication level prior to protocol training | Month 4, Month 8, Month 12, Month 16, Month 20 before training
  Caregivers' assertiveness in communication will be assessed at the beginning of the study using the Cungi and Rey scale. The Cungi and Rey scale is composed of 10 items. The maximum score is 80, the minimum score is 10. A high score reflects a good level of assertiveness in communication.
Caregivers - Evaluate assertiveness in communication | Day 90 after the announcement in the emergency department
  Caregivers' assertiveness in communication will be assessed at the beginning of the study using the Cungi and Rey scale. The Cungi and Rey scale is composed of 10 items. The maximum score is 80, the minimum score is 10. A high score reflects a good level of assertiveness in communication.
Caregivers - Evaluation of self-confidence in complex relational situations addressed during simulation prior to protocol training | Month 4, Month 8, Month 12, Month 16, Month 20 before training
  Caregivers' self-confidence in the complex relational situations addressed during the simulation will be assessed by a self-questionnaire using a Likert-type scale at the start of the study.
Caregivers - Evaluation of self-confidence in complex relational situations addressed during simulation 90 days after training | Day 90 after the announcement in the emergency department
  Caregivers' self-confidence in the complex relational situations addressed during the simulation will be assessed by a self-questionnaire using a Likert-type scale at 90 days after the human simulation training.
Caregivers - Evaluate real-life stress levels in caregivers' professional environment for decision of withholding and withdrawing life-sustaining treatments prior to protocol training | Month 4, Month 8, Month 12, Month 16, Month 20 before training
  Caregivers' stress in their professional environment will be assessed using the Karasek scale, which evaluates mental stress at work at the start of the study. The Karasek scale is composed of 29 items. The maximum score is 116, the minimum score is 29.
Caregivers - Evaluate real-life stress levels in caregivers' professional environment for decision of withholding and withdrawing life-sustaining treatments announcement | Day 90 after the announcement in the emergency department
  Caregivers' stress in their professional environment will be assessed using the Karasek scale, which evaluates mental stress at work at 90 days after human simulation training. The Karasek scale is composed of 29 items. The maximum score is 116, the minimum score is 29.
Caregivers - Evaluating behavior change | Month 4, Month 8, Month 12, Month 16, Month 20 after training
  The theory of behavioural change will be evaluated by a questionnaire completed after training.
Caregivers - Evaluating caregivers' experience of decision of withholding and withdrawing life-sustaining treatments after training | Day 90 after training
  The qualitative evaluation of caregivers' experience of the announcement will be carried out in the form of semi-structured interviews 90 days after the training.
Emergency departments - Implementation of the protocol in practice | Day 90 after training
  The implementation of the protocol will be assessed by the adoption of the announcement protocol by professionals, the deployment of the various components of the intervention protocol (dedicated place, presence of pairs, duration of the announcement, etc.), the adaptations made for announcements of death and decision of withholding and withdrawing life-sustaining treatments. It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.
Emergency departments - Mechanisms of effect of the intervention - Participation and satisfaction of professionals with the training | Day 90 after training
  It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.
Emergency departments - Mechanisms of effect of the intervention - Reactions of families during the LAT | Day 90 after training
  It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.
Emergency departments - Mechanisms of effect of the intervention - Unexpected effects of the use of the announcement protocol | Day 90 after training
  It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.
Emergency departments - Favourable or limiting contextual factors - Departmental organizational factors | Day 90 after training
  It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.
Emergency departments - Favourable or limiting contextual factors - Leadership-facilitator in the team | Day 90 after training
  It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.
Emergency departments - Favourable or limiting contextual factors - Number of emergency department visits with flow analysis | Day 90 after training
  It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.
Emergency departments - Favourable or limiting contextual factors - Characteristics of the patients cared for | Day 90 after training
  It will be evaluated by questionnaires and ad hoc indicators and during semi-structured interviews.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Angers, Angers
  - CH de Bourg-en-Bresse, Bourg-en-Bresse
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Groupement hospitalier centre, Hospices Civils de Lyon, Lyon
  - Groupement hospitalier nord, Hospices Civils de Lyon, Lyon
  - Groupement hospitalier sud, Hospices Civils de Lyon, Lyon
  - CHU de Toulouse, Toulouse
  - CH de Villefranche, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices) may be shared with researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose on request after authorization by the sponsor, the legal department of the Hospices Civils de Lyon and the signature of contract between identified parts.
Supporting Information: Study Protocol
Time Frame: beginning 3 months and ending 5 years following publication
Access Criteria: anne.termoz@chu-lyon.fr

REFERENCES:
- [Derived] Termoz A, Subtil F, Drouin P, Marchal M, Verroul M, Langlois C, Bravant E, Jacquin L, Clement B, Viglino D, Roux-Boniface D, Verbois F, Demarquet M, Dubucs X, Douillet D, Tazarourte K, Schott-Pethelaz AM, Haesebaert J, Douplat M. Evaluating the impact of a standardised intervention for announcing decisions of withholding and withdrawing life-sustaining treatments on the stress of relatives in emergency departments (DISCUSS): protocol for a stepped-wedge randomised controlled trial. BMJ Open. 2024 Sep 5;14(9):e087444. doi: 10.1136/bmjopen-2024-087444. PMID 39237283